CLINICAL TRIAL: NCT05265182
Title: Developing an Immersive Gamification Technology System (ImGTS) for the Management of Patients With Behavioral and Psychological Symptoms of Dementia (Phase 1 Trial)
Brief Title: ImGTS for Patients With Behavioral and Psychological Symptoms of Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augmented eXperience E-health Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: AXEL0001
Record Dates: First submitted 2022-01-14; First posted 2022-03-03 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-07

CONDITIONS: Dementia Alzheimers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: HMD and Semi-Cave
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-CAVE (Experimental): The Semi-CAVE (Figure 2) will use two screens positioned at a corner of the room, each with a ceiling-mounted short throw projector in front. The user will sit in the middle of the area, giving them a viewing angle of roughly 180 degrees. The user will interact with the system through motion sensors positioned at the corners of the area. To one side of the area will be a sufficiently powerful computer running the software. The projectors will be connected to this computer via HDMI cables or similar. The Semi-CAVE may be offered as a solution for rehabilitation centers.
  Interventions: Procedure: virtual reality
- Head-mounted display or HMD (Experimental): The HMD will be a commercially available device that uses handheld controllers in addition to the head mounted apparatus, to control movement while in the VE. This device could provide a cheaper, more practical alternative to patients with mobility issues and environmental limitations brought about by the pandemic, since this can be used at home. Any patient, with supervision from their caregivers, will be able to use the applications using only the HMD system.
  Interventions: Procedure: virtual reality

INTERVENTIONS:
Procedure: virtual reality — Create an immersive technology system for managing the behavioral and psychological symptoms of dementia and determine its acceptability, usability, and safety in the healthy adult population initially, using semi-Cave or head-mounted display.

SUMMARY:
The proposed research project aims to answer the question "Are immersive technology systems effective in the management and treatment of patients with BPSD?". This project is composed of three phases and the current study is the first phase. The phase 1 trial aims to create an immersive technology system for managing the behavioral and psychological symptoms of dementia and determine its acceptability, usability, and safety in the healthy adult population.

DETAILED DESCRIPTION:
The participants will undergo an intervention using the assigned ImGTS for four sessions (twice a week for two weeks), with a maximum of 45 minutes per session. VR trials are in 10- to 20-minute periods with introduction, orientation, and provisions for rest periods for patient comfort. During the experience, documentation of the patient's reaction and interaction with the ImGTS will be recorded by the researchers. The participants will be staying at the designated laboratory for not more than one hour.

Demographic characteristics Demographic characteristics of the participant (age, sex, educational attainment, marital status, living conditions, hobbies and interests, previous experience with VE applications, existing illnesses, medications) will be collected by the researchers through a questionnaire. Personal data, such as name and contact information, will only be collected to allow the investigators to contact the participants, as needed.

Safety Safety will be ensured by assessing a participant's experience of cybersickness. A cybersickness questionnaire, the Virtual Reality Sickness Questionnaire will be administered after each session. In this self-report questionnaire, nine symptoms will be rated as absent/none, slight, moderate, or severe. These symptoms are general discomfort, fatigue, eyestrain, difficulty focusing, headache, fullness of head, blurred vision, dizziness when the eyes are closed, and vertigo. Answering the questionnaire will take around 10 minutes.

In the event that a participant will experience severe cybersickness, they may opt to discontinue the experience. They will be instructed to remove the HMD or to step out of the Semi-CAVE room to rest and recover from the symptoms. A medical professional will be present to monitor the participant's symptoms and to attend to them for further management. The reason(s) for discontinuing the experience will be documented.

Acceptability The acceptability of the design will be measured using the Place Probe, a sense of place questionnaire. The questionnaire will be administered after each session, and it will collect information on a participant's experience in the VE application, particularly on (a) their general impression of the environment, (b) the key features of the environment, and (c) their feelings of presence. A positive general impression, a memorable environment, and high level of presence will indicate that the VE developed is acceptable. This will take about 10 minutes to complete.

Usability Usability testing will be performed according to the PNS ISO/IEC Metrics. The goal is to provide continuous improvement in the design and user experience to maximize the three components of usability: effectiveness, efficiency, and satisfaction. Additional usability metrics will be identified during the first phase of the study. The metrics will be specifically adjusted to the target participants as well as the contents to be included in the VR system.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 to 59 years old
* Montreal Cognitive Assessment-Philippine Version (MoCA-P) score > 20
* Neuropsychiatric Inventory (NPI) score of 0
* Able to understand Filipino and English

Exclusion Criteria:

* Previously diagnosed with dementia
* Receptive aphasia
* Previously diagnosed with a psychiatric disorder
* Previously diagnosed with seizures or epilepsy
* Significant visual and hearing impairment
* Has a history of motion sickness
* Quadriplegia or paralysis of dominant hand
* Life expectancy of less than a year

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
The incidence of cybersickness will be assessed using the Virtual Reality Sickness Questionnaire. | Immediately after each intervention, within an hour of completion of the virtual reality game.
  A 9-item Virtual Reality Sickness Questionnaire to assess cybersickness.
The acceptability of the design will be measured using the Place Probe. | Immediately after each intervention, within an hour of completion of the virtual reality game.
  The Place Probe is a sense of place questionnaire.
The rate of usability will be performed according to the Philippine National Standards ISO/IEC Metrics. | Within an hour of the end of the study.
  The goal is to provide continuous improvement in the design and user experience to maximize the three components of usability: effectiveness, efficiency, and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Veeda Michelle M Anlacan, MD, Principal Investigator — University of the Philippines Manila
Locations (1):
- College of Allied Medical Professions Clinic for Therapy Services, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appel L, Kisonas E, Appel E, Klein J, Bartlett D, Rosenberg J, Smith CN. Administering Virtual Reality Therapy to Manage Behavioral and Psychological Symptoms in Patients With Dementia Admitted to an Acute Care Hospital: Results of a Pilot Study. JMIR Form Res. 2021 Feb 3;5(2):e22406. doi: 10.2196/22406. PMID 33533720
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Birckhead B, Khalil C, Liu X, Conovitz S, Rizzo A, Danovitch I, Bullock K, Spiegel B. Recommendations for Methodology of Virtual Reality Clinical Trials in Health Care by an International Working Group: Iterative Study. JMIR Ment Health. 2019 Jan 31;6(1):e11973. doi: 10.2196/11973. PMID 30702436
- [Background] Clay F, Howett D, FitzGerald J, Fletcher P, Chan D, Price A. Use of Immersive Virtual Reality in the Assessment and Treatment of Alzheimer's Disease: A Systematic Review. J Alzheimers Dis. 2020;75(1):23-43. doi: 10.3233/JAD-191218. PMID 32280091
- [Background] Coelho T, Marques C, Moreira D, Soares M, Portugal P, Marques A, Ferreira AR, Martins S, Fernandes L. Promoting Reminiscences with Virtual Reality Headsets: A Pilot Study with People with Dementia. Int J Environ Res Public Health. 2020 Dec 12;17(24):9301. doi: 10.3390/ijerph17249301. PMID 33322679
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Dominguez JC, Orquiza MG, Soriano JR, Magpantay CD, Esteban RC, Corrales ML, Ampil ER. Adaptation of the Montreal Cognitive Assessment for elderly Filipino patients. East Asian Arch Psychiatry. 2013 Sep;23(3):80-5. PMID 24088400
- [Background] Dominguez J, Fe de Guzman M, Reandelar M, Thi Phung TK. Prevalence of Dementia and Associated Risk Factors: A Population-Based Study in the Philippines. J Alzheimers Dis. 2018;63(3):1065-1073. doi: 10.3233/JAD-180095. PMID 29710725
- [Background] Kales HC, Gitlin LN, Lyketsos CG. Assessment and management of behavioral and psychological symptoms of dementia. BMJ. 2015 Mar 2;350:h369. doi: 10.1136/bmj.h369. PMID 25731881
- [Background] Kim O, Pang Y, Kim JH. The effectiveness of virtual reality for people with mild cognitive impairment or dementia: a meta-analysis. BMC Psychiatry. 2019 Jul 12;19(1):219. doi: 10.1186/s12888-019-2180-x. PMID 31299921
- [Background] Wong WT, Tan NC, Lim JE, Allen JC Jr, Lee WS, Quah JHM, Paulpandi M, Teh TA, Lim SH, Malhotra R. Comparison of Time Taken to Assess Cognitive Function Using a Fully Immersive and Automated Virtual Reality System vs. the Montreal Cognitive Assessment. Front Aging Neurosci. 2021 Nov 23;13:756891. doi: 10.3389/fnagi.2021.756891. eCollection 2021. PMID 34887743
- [Background] Manera V, Chapoulie E, Bourgeois J, Guerchouche R, David R, Ondrej J, Drettakis G, Robert P. A Feasibility Study with Image-Based Rendered Virtual Reality in Patients with Mild Cognitive Impairment and Dementia. PLoS One. 2016 Mar 18;11(3):e0151487. doi: 10.1371/journal.pone.0151487. eCollection 2016. PMID 26990298
- [Background] Mendez MF, Joshi A, Jimenez E. Virtual reality for the assessment of frontotemporal dementia, a feasibility study. Disabil Rehabil Assist Technol. 2015 Mar;10(2):160-4. doi: 10.3109/17483107.2014.889230. Epub 2014 Feb 14. PMID 24524440
- [Background] Moyle W, Jones C, Dwan T, Petrovich T. Effectiveness of a Virtual Reality Forest on People With Dementia: A Mixed Methods Pilot Study. Gerontologist. 2018 May 8;58(3):478-487. doi: 10.1093/geront/gnw270. PMID 28329867
- [Background] Optale G, Urgesi C, Busato V, Marin S, Piron L, Priftis K, Gamberini L, Capodieci S, Bordin A. Controlling memory impairment in elderly adults using virtual reality memory training: a randomized controlled pilot study. Neurorehabil Neural Repair. 2010 May;24(4):348-57. doi: 10.1177/1545968309353328. Epub 2009 Nov 24. PMID 19934445
- [Background] Strong J. Immersive Virtual Reality and Persons with Dementia: A Literature Review. J Gerontol Soc Work. 2020 Apr;63(3):209-226. doi: 10.1080/01634372.2020.1733726. Epub 2020 Feb 24. PMID 32091323
- [Background] Thapa N, Park HJ, Yang JG, Son H, Jang M, Lee J, Kang SW, Park KW, Park H. The Effect of a Virtual Reality-Based Intervention Program on Cognition in Older Adults with Mild Cognitive Impairment: A Randomized Control Trial. J Clin Med. 2020 Apr 29;9(5):1283. doi: 10.3390/jcm9051283. PMID 32365533
- [Background] White PJ, Moussavi Z. Neurocognitive Treatment for a Patient with Alzheimer's Disease Using a Virtual Reality Navigational Environment. J Exp Neurosci. 2016 Nov 8;10:129-135. doi: 10.4137/JEN.S40827. eCollection 2016. PMID 27840579